CLINICAL TRIAL: NCT01506570
Title: A Phase 1 Evaluation of the Safety and Immunogenicity of the Recombinant Live Attenuated Tetravalent Dengue Virus Vaccine Admixtures TV003 and TV005 in Healthy Flavivirus-experienced Adult Subjects
Brief Title: Evaluating the Safety and Immune Response to Two Admixtures of a Tetravalent Dengue Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 280
Record Dates: First submitted 2012-01-05; First posted 2012-01-10 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TetraVax-DV Vaccine - Admixture TV003 (Experimental): Participants will receive one SC injection of the TetraVax-DV Vaccine - Admixture TV003 in their upper arm at Day 0 and Day 180.
  Interventions: Biological: TetraVax-DV Vaccine - Admixture TV003
- TetraVax-DV Vaccine - Admixture TV005 (Experimental): Participants will receive one SC injection of the TetraVax-DV Vaccine - Admixture TV005 in their upper arm at Day 0 and Day 180.
  Interventions: Biological: TetraVax-DV Vaccine - Admixture TV005
- Placebo (Placebo Comparator): Participants will receive one SC injection of placebo in their upper arm at Day 0 and Day 180.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TetraVax-DV Vaccine - Admixture TV003 — One SC injection at Day 0 and Day 180 of the TetraVax-DV Vaccine, Admixture TV003 (10^3 plaque-forming unit [PFU] of rDEN1Δ30, 10^3 PFU of rDEN2/4Δ30[ME], 10^3 PFU of rDEN3Δ30/31-7164, and 10^3 PFU of rDEN4Δ30)
  Arms: TetraVax-DV Vaccine - Admixture TV003
Biological: TetraVax-DV Vaccine - Admixture TV005 — One SC injection at Day 0 and Day 180 of the TetraVax-DV Vaccine, Admixture TV005 (10^3 PFU of rDEN1Δ30, 10^4 PFU of rDEN2/4Δ30[ME], 10^3 PFU of rDEN3Δ30/31-7164, and 10^3 PFU of rDEN4Δ30)
  Arms: TetraVax-DV Vaccine - Admixture TV005
Biological: Placebo — One SC injection at Day 0 and Day 180 of placebo
  Arms: Placebo

SUMMARY:
Dengue viruses can cause dengue fever and other serious health conditions, primarily affecting people living in tropical regions of the world. This study will evaluate the safety and immune responses to two formulations of a tetravalent dengue virus vaccine in healthy adults who have previously been infected with a dengue virus or other flavivirus or have previously received a flavivirus vaccine.

DETAILED DESCRIPTION:
Dengue viruses cause dengue fever and the more severe condition, dengue hemorrhagic fever/shock syndrome. Dengue viruses are common in most tropical and subtropical regions of the world and infection with dengue viruses is the leading cause of hospitalization and death in children in many tropical Asian countries. For these reasons, the World Health Organization (WHO) has made the development of a dengue virus vaccine a top priority. This study will evaluate the safety and immunogenicity of two doses of a live attenuated, tetravalent dengue virus vaccine called TetraVax-DV in healthy adults (18-50 years old) who have previously been infected with a dengue virus or other flavivirus or have previously received a flavivirus vaccine. Two different formulations of the TetraVax-DV vaccine will be evaluated.

Participants will be randomly assigned to receive one of two admixtures of the TetraVax-DV vaccine or a placebo. At a baseline study visit (Day 0), participants will undergo a medical history review, physical examination, blood collection, vital sign measurements, and a pregnancy test for females. Participants will then receive one subcutaneous (SC) injection of their assigned vaccine or placebo in the upper arm. After receiving the vaccine, participants will remain in the clinic for 30 minutes for observation and monitoring. At home, participants will monitor and record their temperature three times a day for 16 days after the first vaccination (from Day 0 through Day 16) and for 16 days after the second vaccination (from Day 180 through Day 196). Additional study visits will occur at Days 3, 8, 10, 12, 14, 16, 21, 28, 56, 90, and 150 and will include a physical examination, vital sign measurements, and blood collection. On Day 180, participants will receive a second SC injection of their assigned vaccine or placebo. Additional study visits will then occur at Days 183, 188, 190, 192, 194, 196, 201, 208, 236, 270, and 360, and will include the same study procedures and monitoring that occurred after the first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* In good general health, as determined by physical examination, laboratory screening, and review of medical history
* Documented history or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus [YFV], St. Louis encephalitis virus [SLE], West Nile virus [WNV], Japanese encephalitis virus [JEV], or tick-borne encephalitis virus [TBEV]) or documented previous receipt of a flavivirus vaccine (licensed or experimental)
* Available for the duration of the study, approximately 26 weeks post-second vaccination
* Willing to participate in the study as evidenced by signing the informed consent document
* Female participants of childbearing potential must be willing to use effective contraception for the duration of the trial. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Currently pregnant, as determined by positive beta-human choriogonadotropin (HCG) test, or breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine, as defined in the protocol
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Any significant alcohol or drug abuse in the 12 months prior to study entry that has caused medical, occupational, or family problems, as indicated by a participant's history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the 6 months prior to study entry)
* HIV infection, by screening and confirmatory assays
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays
* Hepatitis B virus (HBV) infection, by hepatitis B surface antigen (HBsAg) screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 42 days following vaccination
* Asplenia
* Receipt of blood products within the 6 months prior to study entry, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 42 days following vaccination
* Anticipated receipt of any investigational agent in the 42 days before or after vaccination
* Has definite plans to travel to a dengue endemic area during the study
* Refusal to allow storage of specimens for future research

Additional Inclusion Criteria for Second Dose of Vaccine:

* In good general health, as determined by physical examination and review of medical history
* Available for the duration of the study, approximately 6 months post-vaccination
* Female participants of childbearing potential must be willing to use effective contraception for the duration of the trial. More information on this criterion can be found in the protocol.

Exclusion Criteria for Second Dose of Vaccine:

* Anaphylaxis or angioedema following the first dose of vaccine
* Currently pregnant, as determined by positive beta-HCG test, or breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Any significant alcohol or drug abuse in the 12 months prior to study entry that has caused medical, occupational, or family problems, as indicated by a participant's history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the 6 months prior to study entry)
* HIV infection, by screening and confirmatory assays
* HCV infection, by screening and confirmatory assays
* HBV infection, by HBsAg screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 42 days following vaccination
* Asplenia
* Receipt of blood products within the 6 months prior to study entry, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 42 days following vaccination
* Anticipated receipt of any other investigational agent in the 42 days before or after vaccination
* Has definite plans to travel to a dengue endemic area during the study
* Refusal to allow storage of specimens for future research

Other Treatments and Ongoing Exclusion Criteria:

The following criteria will be reviewed on Days 28 and 56 following each vaccination. If any become applicable during the study, the participant will not be included in further immunogenicity evaluations, as of the exclusionary visit. The participant will, however, be encouraged to remain in the study for safety evaluations for the duration of the study.

Ongoing Exclusion Criteria:

* Use of any investigational drug or investigational vaccine other than the study vaccine during the 42-day period post-vaccination
* Chronic administration (greater than or equal to 14 days) of steroids (defined as prednisone equivalent of greater than or equal to 10 mg per day), immunosuppressants, or other immune-modifying drugs initiated during the 42-day period post-vaccination (topical and nasal steroids are allowed)
* Receipt of a licensed vaccine during the 42-day period post-vaccination
* Receipt of immunoglobulins and/or any blood products during the 42-day period post-vaccination
* Pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2011-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Safety of TetraVax-DV TV003 and TV005, as assessed by the frequency of vaccine-related adverse events | Measured through Day 360
Immunogenicity of TV003 and TV005, as assessed by neutralizing antibody titers to DENV-1, DENV-2, DENV-3, and DENV-4 | Measured 28, 56, 90, and 180 days after each vaccination
  Monovalent, bivalent, trivalent, and tetravalent seropositivity rates will be determined at 28, 56, and 90 days after each vaccination.
Whether a second dose of the vaccine given at Day 180 will induce seropositivity in those participants that remained seronegative to one or more DENV serotypes following the first vaccination | Measured through Day 360

SECONDARY OUTCOMES:
Frequency, quantity, and duration of viremia following vaccination | Measured through Day 360
Number of flavivirus-experienced vaccinees infected with DENV-1, DENV-2, DENV-3, and DENV-4 | Measured through Day 360
  Infection is defined as recovery of vaccine virus from the blood or serum of a participant and/or by developing seropositivity to DEN virus (plaque reduction neutralization titer [PRNT]50 greater than or equal to 1:10).
Duration of the neutralizing antibody response | Measured 26 weeks after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Locations (3):
- United States (3):
  - Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland
  - Fletcher Allen Health Care (FAHC), General Clinical Research Center (GCRC), Burlington, Vermont
  - University of Vermont Vaccine Testing Center, Burlington, Vermont

REFERENCES:
- [Background] Bhamarapravati N, Sutee Y. Live attenuated tetravalent dengue vaccine. Vaccine. 2000 May 26;18 Suppl 2:44-7. doi: 10.1016/s0264-410x(00)00040-2. PMID 10821973
- [Background] Blaney JE Jr, Durbin AP, Murphy BR, Whitehead SS. Development of a live attenuated dengue virus vaccine using reverse genetics. Viral Immunol. 2006 Spring;19(1):10-32. doi: 10.1089/vim.2006.19.10. PMID 16553547
- [Background] Durbin AP, Kirkpatrick BD, Pierce KK, Schmidt AC, Whitehead SS. Development and clinical evaluation of multiple investigational monovalent DENV vaccines to identify components for inclusion in a live attenuated tetravalent DENV vaccine. Vaccine. 2011 Sep 23;29(42):7242-50. doi: 10.1016/j.vaccine.2011.07.023. Epub 2011 Jul 21. PMID 21781997
- [Derived] Whitehead SS, Durbin AP, Pierce KK, Elwood D, McElvany BD, Fraser EA, Carmolli MP, Tibery CM, Hynes NA, Jo M, Lovchik JM, Larsson CJ, Doty EA, Dickson DM, Luke CJ, Subbarao K, Diehl SA, Kirkpatrick BD. In a randomized trial, the live attenuated tetravalent dengue vaccine TV003 is well-tolerated and highly immunogenic in subjects with flavivirus exposure prior to vaccination. PLoS Negl Trop Dis. 2017 May 8;11(5):e0005584. doi: 10.1371/journal.pntd.0005584. eCollection 2017 May. PMID 28481883